CLINICAL TRIAL: NCT03991975
Title: Phase Ib Study to Evaluate the Safety and Efficacy of TQB2450 (PD-L1 Antibody) Combined With Anlotinib in Subjects With Advanced Acral Malignant Melanoma
Brief Title: Study of TQB2450 Combined With Anlotinib in Subjects With Advanced Acral Malignant Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-09
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-01

CONDITIONS: Advanced Acral Malignant Melanoma
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib + TQB2450 (Experimental): TQB2450 1200 mg IV on Day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycles (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: Anlotinib; Drug: TQB2450

INTERVENTIONS:
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor.
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

SUMMARY:
TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.

ELIGIBILITY:
Inclusion Criteria:

1.18 and 75 years; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

2. Histologically or cytologically confirmed advanced acral malignant melanoma. 3. At least one measurable lesion. 4. Providing tumor specimen obtained by biopsy or surgical sample within 2 years.

5. Has received at least first-line treatment but appeared disease progression or intolerance.

6. The main organs function are normally, the following criteria are met:

1. hemoglobin ≥ 90 g/L; neutrophils ≥ 1.5*10^9/L; platelets ≥ 100 x 10^9/ L;
2. total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN ; serum creatinine ≤1╳ULN，creatinine clearance >50 umol/L ;
3. INR, aPTT, PT≤1.5 x ULN;
4. left ventricular ejection fraction (LVEF) ≥50%. 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

8.Understood and signed an informed consent form.

Exclusion Criteria:

1. Prior therapy with VEGFR-target TKI included anlotinib or an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody ,or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
2. Hypersensitivity to recombinant humanized anti-PD-1 monoclonal Abm or its components.
3. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix.
4. Has any active autoimmune disease or history of autoimmune disease.
5. Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration.
6. Has multiple factors affecting oral medication.
7. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
8. Has any bleeding or bleeding events ≥ grade 3 or with unhealed wounds, ulcerative , or fractures within 4 weeks prior to the first administration.
9. Has uncontrollable symptoms of brain metastasis, spinal cord compression, cancerous meningitis during screening within 8 weeks before first dose.
10. Has received chemotherapy, surgery, radiotherapy, the last treatment from the first dose less than 4 weeks, or oral targeted drugs for less than 5 half-lives, or oral fluorouracil pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks.
11. Has any serious and / or uncontrolled disease.
12. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first dose.
13. Has received granulocyte colony stimulating factor(G -CSF)，or Granulocyte macrophage colony stimulating factor (GM-CSF) within 4 weeks prior to first dose.
14. According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases including mental disorders need to be treated together, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 21 days
  Maximum tolerated dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) of Anlotinib and TQB2450 in advanced acral malignant melanoma patients, Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-21).
Maximum tolerated dose (MTD) | up to 21 days
  MTD defined as the highest dose level at which less than or equal to 2 of 6 subjects experience dose limiting toxicity (DLT)
Recommended Phase II dose (RP2D) | up to 24 months
  The RP2D defined as the lower dose level to MTD based on the safety profile
Overall response rate (ORR) | up to 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD)
Progression-free survival (PFS) | up to 24 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause
Overall survival (OS) | up to 24 months
  OS defined as the time from randomization to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive
Adverse Event | up to 24 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijin, Beijing Municipality, China

REFERENCES:
- [Derived] Du Y, Dai J, Mao L, Wei X, Bai X, Chen L, Lin J, Chi Z, Cui C, Sheng X, Lian B, Tang B, Wang X, Yan X, Li S, Zhou L, Guo J, Chen Y, Si L. Phase Ib study of anlotinib in combination with anti-PD-L1 antibody (TQB2450) in patients with advanced acral melanoma. J Eur Acad Dermatol Venereol. 2024 Jan;38(1):93-101. doi: 10.1111/jdv.19467. Epub 2023 Sep 4. PMID 37625814